CLINICAL TRIAL: NCT06883370
Title: Analgesic Evaluation of Ultrasound Guided Transversalis Fascia Plane (Tfp) Block With 0.4 ml/kg of Ropivacaine 0.375 % in Paediatric Laparoscopic Inguinal Hernia Repair.
Brief Title: Analgesia Evaluation of an Ultrasound-guided Technique for Inguinal Hernia Surgery in Children in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JEPUKM-JEP-2023-518
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Inguinal Hernia; Surgery; Paediatric
Keywords: Ultrasound; transversalis fascia; ropivacaine; inguinal hernia; paediatric patients
MeSH Terms: conditions — Hernia, Inguinal | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients (Experimental): All paediatric patients undergoing inguinal hernia repair
  Interventions: Combination Product: ultrasound-guided transversals fascia plane block with ropivacaine

INTERVENTIONS:
Combination Product: ultrasound-guided transversals fascia plane block with ropivacaine — using 0.375% ropivacaine of 0.4mls/kg

SUMMARY:
The basis for the transversalis fascia plane (TFP) block involves infiltration of local anaesthetic blocking the ilioinguinal and iliohypogastric nerve which are located between the fascia of the transversus abdominis muscle and the transversalis fascia. The fascia of the transversus abdominis muscle, also called the thoracolumbar fascia, is formed when the transversus abdominis and internal oblique muscles taper off posteriorly into a common aponeurosis and abuts the lateral border of quadratus lumborum muscle. The transversalis fascia is a thin aponeurotic membrane which lies between the transversus abdominis muscle and the extraperitoneal fascia, and is part of the general layer of fascia lining the abdominal cavity. Thus the TFP block is said to be suitable for lower abdominal surgery.

This study was designed obtain the analgesic efficacy of ropivacaine 0.375% for ultrasound-guided (USG) TFP block for paediatric patients undergoing laparoscopic inguinal hernia.

DETAILED DESCRIPTION:
Methods: Thirty-two ASA 1 or 2 patients, aged 6 months to 12 years old undergoing laparoscopic inguinal hernia repair were recruited into this study. They were all given 0.4ml/kg of ropivacaine 0.375% after induction of anaesthesia. Intra operative heart rate (HR), mean arterial pressure (MAP), cumulative fentanyl consumption as well as post operative FLACC score, post operative nausea and vomiting incidence, time to first oral intake, parental satisfaction and complications were recorded.

ELIGIBILITY:
Inclusion Criteria: All ASA I or II patients undergoing inguinal hernia repair

Exclusion Criteria: Parent's refusal, allergic to study drug

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of ultrasound-guided transversals fascia plane block in paediatric | immediate post operative
  Pain score

CONTACTS AND LOCATIONS:
Overall Officials: Dr, Principal Investigator — The National University of Malaysia
Locations (1):
- The National University of Malaysia, Kuala Lumpur, Malaysia